CLINICAL TRIAL: NCT03867344
Title: The Functional Neuroanatomy of the Human Physiological Stress Response
Acronym: Hypo fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Boston Children's Hospital (Other); Mclean Hospital (Other)
Responsible Party: Principal Investigator, Gail Kurr Adler, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019P000318
Record Dates: First submitted 2019-03-04; First posted 2019-03-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hypoglycemia; Physiological Stress
Keywords: Hypoglycemia; Stress; Brain
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoglycemia (Active Comparator): Participants undergo Autonomic Nervous System (ANS) Testing (measurement of Baroreflex Sensitivity using the Modified Oxford test) followed by a functional MRI (fMRI) scan. The next day, participants undergo one 120-minute hypoglycemic hyperinsulinemic clamp procedure (50mg/dL) in the morning followed by ANS Testing and an fMRI scan. Four days later, participants undergo repeat ANS Testing and an fMRI scan.
  Interventions: Other: Hypoglycemic Hyperinsulinemic Clamp
- Normoglycemia (Placebo Comparator): Participants undergo Autonomic Nervous System (ANS) Testing (measurement of Baroreflex Sensitivity using the Modified Oxford test) followed by a functional MRI (fMRI) scan. The next day, participants undergo one 120-minute normoglycemic hyperinsulinemic clamp procedure (90mg/dL) in the morning followed by ANS Testing and an fMRI scan. Four days later, participants undergo repeat ANS Testing and an fMRI scan.
  Interventions: Other: Normoglycemic Hyperinsulinemic Clamp

INTERVENTIONS:
Other: Hypoglycemic Hyperinsulinemic Clamp — Participants undergo a 120-minute hypoglycemic hyperinsulinemic clamp procedure.
  Other Names: Hypoglycemic Hyperinsulinemic Clamp Procedure
  Arms: Hypoglycemia
Other: Normoglycemic Hyperinsulinemic Clamp — Participants undergo a 120-minute normoglycemic hyperinsulinemic clamp procedure.
  Other Names: Normoglycemic Hyperinsulinemic Clamp Procedure
  Arms: Normoglycemia

SUMMARY:
The purpose of this study is to examine the effect of a moderately low blood sugar stress on the nervous system. The investigators hope that information obtained from completing this study will help to reveal information about how a non-psychological stress impacts the parts of the brain that react to stress and the autonomic nervous system. The autonomic nervous system is the part of the nervous system that provides the body with involuntary or automatic control of heart rate, blood pressure, and breathing.

DETAILED DESCRIPTION:
Stress is common in daily life and is associated with adverse health outcomes. This proposal will study how a physiological stress (low blood sugar), a stress often experienced by people with diabetes, affects connections in the brain. The investigators will focus on brain connections that are involved in autonomic control of cardiovascular function, and determine both how these brain connections are altered by low blood sugar and how these alterations associate with changes in pain perception and cardiovascular control.

In this study, the investigators introduce a novel mechanistic, integrative approach to the assessment of the response to and recovery from a specific physiologic stressor - insulin-induced hypoglycemia. The overall hypothesis is that a hypoglycemic stress will alter autonomic brain networks, and will affect clinically relevant physiological outcomes (cardiovascular autonomic function); and that the rate and extent of recovery of these brain networks will provide a measure of resilience.

In combination, this approach will allow the investigators for the first time to define the magnitude of the effect of stress exposure on neural circuitry and on clinically relevant stress-related physiological outcomes (cardiovascular autonomic function) and to define the recovery of brain circuitry and these related physiological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Males and Females age 18 to 45 years
* BMI 18-35 kg/m2

Exclusion Criteria:

* Pregnancy
* Lactation
* Menopause
* Any medical condition
* Current or prior alcohol or drug abuse
* Active tobacco use
* Abnormal ECG
* In all subjects, any individuals on oral, injected, inhaled or topical corticosteroids within the last year or oral contraceptives within the past 3 months will be excluded.
* Use of medications other than thyroid hormone or hormonal birth control
* Serum potassium >5.0 mmol/L
* Estimated GFR <60 mL/min/1.73 m2
* Hemoglobin A1c ≥6.5%
* Patient Health Questionnaire (PHQ9) for depression score ≥15
* GAD-7 Questionnaire for anxiety score ≥10
* PTSD Checklist for DSM-5 (PCL-5) score ≥31
* Perceived Stress Scale (PSS-14) score >28
* Blood pressure systolic ≥140 or <100 mmHg; Blood pressure diastolic >90 mmHg
* Metal in the body including: cardiac pacemakers, stents, artificial heart valves, artificial limbs or hands, brain stimulator devices, implanted drug pumps, ear implants, eye implants or known metal fragments in eyes, exposure to shrapnel or metal filings (wounded in military combat, sheet metal workers, welders, and others), other metallic surgical hardware in vital areas, certain tattoos with metallic ink, certain transdermal medication patches, and metal-containing IUDs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Effect of physiological stress (hypoglycemia) on brain networks involved in autonomic function | Baseline, 8 hours after physiological stress, and 4 days after physiological stress
  Functional MRI will be performed following physiological stress (hypoglycemia) or placebo (normoglycemia) and a functional connectivity analysis will be performed on the fMRI data. The outcome will be alterations in neural network connectivity, as measured by changes in Pearson-correlation coefficients among the following brain structures: right anterior insula and anterior cingulate cortex; right anterior insula and hypothalamus; hypothalamus and anterior cingulate cortex; hypothalamus and amygdala; locus coeruleus and hypothalamus.
The relationship over time between stress-induced changes in brain networks and stress-induced changes in baroreflex sensitivity | Baseline, 8 hours after physiological stress, and 4 days after physiological stress
  The stress-induced change in baroreflex sensitivity (msec/mmHg) will be determined. Pearson correlation coefficients (r) between the changes in baroreflex sensitivity and the changes in brain connectivity (right anterior insula and anterior cingulate cortex; hypothalamus and amygdala [determined for the first outcome above]) will be calculated and tested for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital; David Borsook, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The data collected will comply with the NIH requirements for timely release and data sharing. Data will be shared in the form of publications and presentations in scientific forums. As the NIH has noted, the investigators reserve the right to keep the data restricted in order to perform the initial analyses for this grant proposal and will continue to use the data for further, but not prolonged, exclusive use. Of note, the sharing of this data will be limited by at least the following issues, some unique to this proposal and some not unique. Some of the data obtained in this study is defined to be sensitive in nature, which may restrict its ability to be shared. Data may only be shared with the approval of our IRB and is limited by HIPPA and any other regulations that may be promulgated during the course of this proposal.
Time Frame: Data will be shared after completion of study and initial publications which we anticipate to be within 18 months of the final participant completing the study protocol.
Access Criteria: Access to data must be approved by the IRB at our institution.